CLINICAL TRIAL: NCT05285358
Title: Safety of Pressurized Intraperitoneal Aerosolized Chemotherapy (PIPAC) in Biliary Tract Cancer Patients With Peritoneal Metastases
Brief Title: Pressurized Intraperitoneal Aerosolized Nab-Paclitaxel in Combination With Gemcitabine and Cisplatin for the Treatment of Biliary Tract Cancer Patients With Peritoneal Metastases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21679; NCI-2022-01766 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21679 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Distal Bile Duct Adenocarcinoma; Gallbladder Carcinoma; Intrahepatic Cholangiocarcinoma; Metastatic Malignant Neoplasm in the Peritoneum; Stage IV Distal Bile Duct Cancer AJCC v8; Stage IV Intrahepatic Bile Duct Cancer AJCC v8; Stage IV Intrahepatic Cholangiocarcinoma AJCC v8; Stage IVB Gallbladder Cancer AJCC v8
MeSH Terms: conditions — Gallbladder Neoplasms; Cholangiocarcinoma | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (gemcitabine, cisplatin, nab-paclitaxel PIPAC) (Experimental): Patients receive gemcitabine IV over 30 minutes and cisplatin IV over 60 minutes on days 1 and 8. Patients also receive nab-paclitaxel via PIPAC over 5-10 minutes on day 3 of cycles 1, 3, and 5. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Drug: Nab-paclitaxel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Drug: Nab-paclitaxel — Given via PIPAC
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; Protein-bound Paclitaxel
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial studies the side effects of pressurized intraperitoneal aerosolized chemotherapy (PIPAC) nab-paclitaxel in combination with gemcitabine and cisplatin in treating patients with biliary tract cancer that has spread to the peritoneum (peritoneal metastases). PIPAC involves the administration of intraperitoneal chemotherapy (anticancer drugs given directly to the lining of the abdomen). PIPAC uses a nebulizer (a device that turns liquids into a fine mist) which is connected to a high-pressure injector and inserted into the abdomen (part of the body that contains the digestive organs) during a laparoscopic procedure (a surgery using small incisions to introduce air and insert a camera and other instruments into the abdominal cavity for diagnosis and/or to perform routine surgical procedures). Pressurization of the liquid chemotherapy through the study device results in aerosolization (a fine mist or spray) of the chemotherapy intra-abdominally (into the abdomen), which results in the drug reaching more of the tissue as well as reaching deeper into the tissue, which reduces the amount of chemotherapy that needs to be used and potentially reduces side effect. Chemotherapy drugs, such as nab-paclitaxel, gemcitabine, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving nab-paclitaxel via PIPAC in combination with standard of care gemcitabine and cisplatin may reduce side effects and make this chemotherapy regimen more tolerable in patients with biliary tract cancer that has spread to the spread to the peritoneum.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the safety of PIPAC nab-paclitaxel in combination with systemic chemotherapy in patients with biliary tract cancer with peritoneal metastases, based on treatment-related adverse events reported by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OBJECTIVES:

I. Efficacy. II. Post-operative surgical complications by Clavien-Dindo classification evaluated at 4 weeks after each PIPAC.

III. Median overall survival and median progression-free survival. IV. PIPAC technical failure rate. V. Patient-reported health state/quality of life and symptoms before treatment (week 1) and at weeks 7, 13, 19, and 25/off study, as measured by the European Quality of Life Five Dimension Five Level Scale Questionnaire (EQ-5D-5L) and MD Anderson Symptom Inventory (MDASI).

VI. Functional status, as measured by the number of daily steps before and after treatments (Vivofit 4 wristband pedometer - Garmin Company).

EXPLORATORY OBJECTIVES:

I. Characterization of sub-clonal evolution and tumor microenvironment in response to therapy with a particular focus on immune subsets.

II. Pharmacokinetic and pharmacodynamic evaluations to evaluate the therapeutic advantage of PIPAC nab-paclitaxel delivery.

OUTLINE:

Patients receive gemcitabine intravenously (IV) over 30 minutes and cisplatin IV over 60 minutes on days 1 and 8. Patients also receive nab-paclitaxel via PIPAC over 5-10 minutes on day 3 of cycles 1, 3, and 5. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Age: >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histologically or cytologically confirmed intrahepatic cholangiocarcinoma or extrahepatic cholangiocarcinoma or gallbladder cancer
* Documented metastatic disease on computed tomography (CT) imaging or magnetic resonance imaging (MRI). CT scan or MRI to assess measurable disease must have been completed within 28 days prior to registration
* Visible peritoneal metastatic disease on cross-sectional imaging or diagnostic laparoscopy (does not have to be measurable by Response Evaluation Criteria in Solid Tumors [RECIST] 1.1)
* Fully recovered from acute toxic effects (except alopecia, hearing loss, or non-clinically significant laboratory abnormalities) =< grade 1 of prior anti-cancer therapy
* Complete medical history and physical exam (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)
* Absolute neutrophil count (ANC) >= 1,500/mcL (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)
* Platelets >= 100,000/mcL (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)
* Hemoglobin >= 8 g/dL (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)
* Serum albumin >= 2.8 g/dL (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)
* Total bilirubin =< 1.5 X upper limit of normal (ULN) (unless has Gilbert's disease, then direct bilirubin < 1.5 mg/dL) (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)
* Aspartate aminotransferase (AST) =< 5 x ULN (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)
* Alanine aminotransferase (ALT) =< 5 x ULN (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)
* Calculated creatinine clearance of >= 45 mL/min per 24 hour urine test or the Cockcroft-Gault formula (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)
* Seronegative for human immunodeficiency virus (HIV) antigen (Ag)/antibody (Ab) combo (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)

  * If seropositive, patient may be eligible if they are stable on antiretroviral therapy, have a CD4 T cell count >= 200/µL, and have an undetectable viral load
* Documented virology status of hepatitis, confirmed by hepatitis B virus (HBV) and hepatitis C virus (HCV) tests (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)

  * For patients with active HBV, HBV deoxyribonucleic acid (DNA) < 500 IU/mL during screening, initiation of anti-HBV treatment at least 14 days prior to day 1 of cycle 1, and willingness to continue anti-HBV treatment during the study (per standard of care)
  * If seropositive for HCV, nucleic acid quantification must be performed. Viral load must be undetectable
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated)

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential* to use an effective method of birth control (e.g. licensed hormonal/barrier methods or surgery intended to prevent pregnancy [or with a side effect of pregnancy prevention]) or abstain from heterosexual activity for the course of the study through at least 14 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Any prior systemic therapy treatment for advanced cholangiocarcinoma or gallbladder cancer
* Any prior adjuvant therapy (chemotherapy, radiation therapy, biological therapy, immunotherapy) completed < 6 months prior to registration
* Strong CYP3A4 inducers/inhibitors within 14 days prior to day 1 of protocol therapy
* Bowel obstruction requiring nasogastric tube, percutaneous endoscopic gastrostomy, or exclusive total parenteral nutrition
* Evidence of liver metastases with >= 50% liver occupation
* Any history of, or current, brain or subdural metastases
* Life expectancy < 3 months
* History of peripheral neuropathy >= grade 2 measured by NCI CTCAE version 5.0 ("moderate symptoms, limiting instrumental activities of daily living")
* Treatment with therapeutic oral or IV antibiotics within 14 days prior to day 1 cycle 1 of treatment

  * Patients receiving prophylactic antibiotics are eligible, provided the signs of active infection have resolved
* Any prior malignancy except adequately treated basal or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for two years
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agents (platinum-based compounds, etc.)
* Clinically significant uncontrolled illness
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2028-10-11 (Estimated); Study Completion 2028-10-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 6 weeks after cycle 1 (1 cycle = 21 days)
  Measured by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Toxicities observed during the first 6 weeks after the first cycle will be summarized by type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study treatment, and reversibility or outcome.

SECONDARY OUTCOMES:
Efficacy - RECIST | Up to 1 year after completion of chemotherapy
  Measured by Response Evaluation Criteria in Solid Tumors (RECIST) via computerized tomography (CT) scan.
Efficacy - PGRS | Up to 1 year after completion of chemotherapy
  Measured by Peritoneal Regression Grading Score (PGRS) via biopsy at each Pressurized Intraperitoneal Aerosolized Chemotherapy (PIPAC) cycle.
Efficacy - PCI | Up to 1 year after completion of chemotherapy
  Measured by Peritoneal Carcinomatosis Index (PCI) at the time of laproscopy.
Post-operative surgical complications | Up to 4 weeks after each pressurized intraperitoneal aerosolized chemotherapy treatment
  Measured by Clavien-Dindo classification. Results will be strictly descriptive in nature.
Overall survival | From initiation of treatment to death, assessed up to 1 year
  The length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive.
Progression-free survival | From initiation of treatment to progression, assessed up to 1 year
  Will be described using the Kaplan-Meier method.
Change in patient-reported health state/quality of life and symptoms | Before treatment (week 1) up to 1 year
  Measured by the European Quality of Life Five Dimension Five Level Scale Questionnaire and MD Anderson Symptom Inventory.
Functional status | Up to 1 year
  Measured by the number of daily steps before and after treatments (Vivofit 4 wristband pedometer - Garmin Company).

CONTACTS AND LOCATIONS:
Overall Officials: Daneng Li, MD, Principal Investigator — City of Hope Medical Center; Mustafa Raoof, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Li D, Crook C, Chung V, Brar G, Fakih M, Barzi A, Melstrom L, Singh G, Fong Y, Frankel P, Raoof M. Safety of pressurized intraperitoneal aerosolized chemotherapy in biliary cancer patients with peritoneal metastases. Future Oncol. 2024;20(33):2521-2531. doi: 10.1080/14796694.2024.2394013. Epub 2024 Sep 12. PMID 39263892